CLINICAL TRIAL: NCT02116647
Title: Role of Psychoanalysis in Prevention of Girl Child Maltreatment and Neglect: A Randomized Controlled Trial
Brief Title: Role of Psychoanalysis in Prevention of Girl Child Maltreatment and Neglect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Macmillan Research Group UK (Industry)
Collaborators: Sonal Foundation, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Mac/NMP 1130
Record Dates: First submitted 2014-04-15; First posted 2014-04-17 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2014-07

CONDITIONS: Abuse Neglect; Social; Deprivation, Maltreatment Syndrome (Infant or Child)
Keywords: Gender discrimination; Psychoanalysis; Randomized controlled trial
MeSH Terms: conditions — Sexism | interventions — Psychoanalytic Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Psychoanalytic therapy (Experimental): manualized psychoanalytic psychotherapy
  Interventions: Behavioral: Psychoanalytic therapy
- Control Group (No Intervention): Standard care

INTERVENTIONS:
Behavioral: Psychoanalytic therapy
  Arms: Psychoanalytic therapy

SUMMARY:
In India, precisely northern states, skewed sex ratios, female feticide and higher child mortality rates for girls have become serious concern. The female child mortality as a result of son preference have increased during the last several decades .Since families cannot know the sex of the fetus due to Indian government policies, maltreatment and serious neglect has been tools to ensure there are few survivors.

ELIGIBILITY:
Inclusion Criteria:

* Families having girl child before
* High risk families with high expectation of having son

Exclusion Criteria:

* Families having son before
* Relocation and moving out of town during study period
* Not ready to consent for intervention

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 134 (Actual)
Dates: Start 2012-11; Primary Completion 2013-08 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Post Natal Depression | Change from baseline in Edinburgh Postnatal Depression Scale at 6 weeks

SECONDARY OUTCOMES:
Mother-infant interaction | Change from Baseline in Parent/Caregiver Involvement Scale at 6 weeks

OTHER OUTCOMES:
Abuse and neglect outcomes | Upto six weeks reported incidences of abuse and maltreatment

CONTACTS AND LOCATIONS:
Overall Officials: Bharat Chaudhari, MA, Study Director — Sonal Foundation, India; Mandy Conlon, MA, Study Chair — Goldington Family Center, UK
Locations (2):
- India (2):
  - Sonal Foundation, Ahmedabad, Gujarat
  - NMP Medical Research Institute, Jhunjhunūn, Rajasthan